CLINICAL TRIAL: NCT00515840
Title: GPIAG and Leicester Asthma and Dysfunctional Breathing (GLAD) Study: a Randomised Controlled Study
Acronym: GLAD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: P Burns (Other)
Collaborators: University Hospitals, Leicester (Other)
Responsible Party: Sponsor-Investigator, P Burns, Research Governance Manager, University of Aberdeen
Organization: University of Aberdeen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03/014
Record Dates: First submitted 2007-08-13; First posted 2007-08-14 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Asthma; Respiratory
MeSH Terms: conditions — Asthma | interventions — Physical Therapists

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Sham Comparator): equal time with health care professional (asthma nurse)
  Interventions: Other: Physiotherapist

INTERVENTIONS:
Other: Physiotherapist — Physiotherapist administered breathing retraining programme

SUMMARY:
Breathing retraining supervised by a physiotherapist will result in improvements in the quality of life and asthma control of patients treated for asthma in the community with symptoms suggestive of dysfunctional breathing.

To investigate the effects of breathing retraining on clinical and physiological parameters of asthma control, to identify the characteristics of patients who benefit, to perform a health economic evaluation.

DETAILED DESCRIPTION:
Objectives:

* To assess the effect of breathing retraining on asthma-related health status, asthma control and objective indices of asthma severity (bronchial hyper-reactivity (BHR), sputum eosinophilia and nitric oxide production) in patients with symptomatic asthma.
* To compare the relationship between symptoms of dysfunctional breathing (Nijmegen Questionnaire screening score), changes in asthma-related health status and other parameters resulting from breathing retraining
* To explore the relationship between dysfunctional breathing, baseline asthma symptoms, treatment and asthma-related quality of life.
* To estimate the cost effectiveness of the breathing retraining intervention

ELIGIBILITY:
Inclusion Criteria:

* Asthma diagnosis in medical records
* Age 17-70 yrs.
* One or more prescription for asthma medication in previous 12 months
* Impaired asthma related quality of life (AQLQ score <5.5)

Exclusion Criteria:

* COPD
* Unstable or under-treated asthma at enrollment.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2003-10; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Change in AQLQ scores between intervention and control groups in subjects with positive NQ screening scores 1 month post intervention Change in AQLQ scores between intervention groups of subjects with positive and negative NQ screening scores | Dec 2006

SECONDARY OUTCOMES:
Changes in bronchial hyperresponsiveness(PC 20), sputum eosinophil counts and exhaled NO between intervention and control groups in subjects with positive and negative NQ screening scores Change in ACQ Score between the intervention and the control gr | Dec 2007

CONTACTS AND LOCATIONS:
Overall Officials: Mike Thomas, Principal Investigator — University of Aberdeen